CLINICAL TRIAL: NCT02644928
Title: Effects of Weight Loss on Renal Function in Obese Patients With Chronic Kidney Disease Undergoing Bariatric Surgery
Brief Title: Weight Loss in Obese Kidney Disease Patients After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Enrique Morales Ruiz, MD (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, Enrique Morales Ruiz, MD, Principal Investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Other Study IDs: HDOC-BAROBE-2015-01
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Disease; Bariatric Surgery Candidate
Keywords: Chronic kidney disease; Bariatric Surgery Candidate; Caloric restriction
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — In this study, blood and urine samples will be collected to determine the effect of weight loss in proteinuria and renal function.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed as a prospective, single-center, longitudinal and analytical study on the effect of bariatric surgery in obese patients with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
It is expected to enroll 22 obese subjects with chronic kidney disease (decrease in glomerular filtration and/or albuminuria/proteinuria). After the inclusion in the study patients will remain for six months with a reduced calorie diet until the day of bariatric surgery. Time monitoring of the patient after surgery is 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years (male or female).
* BMI >35 kg/m2 who meet the following criteria:

  1. GFR 30-60 ml/min and proteinuria>1g/24 hours despite receiving maximally tolerated doses of blocking the renin-angiotensin system.
  2. GFR >60 ml/min and proteinuria >(3.5) 2.5 g/24 hours despite receiving maximally tolerated doses of blocking the renin-angiotensin system.
* Patients with BMI> 40 kg/m2 with a GFR> 30 ml/min and proteinuria >(1) 0.5 g/24 hours despite receiving maximally tolerated doses of blocking the renin-angiotensin system.
* Patients who are able to understand the purpose and risks of the study, which has been fully informed and have finally given the written informed consent according to the ICH-GCP. Patients who can not read or write but who properly understand the verbal information provided by the investigator (or sub-investigator) the consent will be granted orally before their inclusion and an independent witness will signing the informed consent document.

Exclusion Criteria:

* Subjects who are participating or have participated in another clinical trial and/or who are taking or have taken an experimental drug (not registered) in the last 28 days.
* Patients with chronic renal replacement therapy (hemodialysis and/or peritoneal dialysis) and/or renal transplantation.
* Patients with poorly controlled blood pressure (SBP> 170 mmHg or DBP> 110 mmHg).
* Patients with a history of cardiovascular events (stroke, ischemic heart disease) in the past six months.
* Patients treated with steroids or other immunosuppressants.
* Patients with a history of renovascular disease, obstructive uropathy, autoimmune diseases, cancer, drug use.
* Patients who are pregnant or lactating.
* Patients who do not sign the informed consent.
* A slight chance of compliance with visits scheduled in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese subjects with renal pathology (decrease in glomerular filtration and/or albuminuria/proteinuria) who are candidates to bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Reduction of proteinuria/albuminuria in patients with obesity and nephropathy of any etiology treated with bariatric surgery | 24 months
  Reduction (measured as a percentage) of proteinuria/albuminuria in patients with obesity after bariatric surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Morales Ruiz, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No